CLINICAL TRIAL: NCT00172640
Title: Identification of Differentially Expressed Genes in Hepatocellular Carcinoma With DNA Microarrays
Brief Title: Genetic Studies in Liver Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Industrial Technology Research Institute, Taiwan (Other)
Other Study IDs: 9361701211
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Hepatocellular carcinoma (HCC) is one the most common malignancies in the world, especially in sub-Saharan Africa and Southeast Asia. Since 1984, it has been the leading cause of cancer death in Taiwan. About 6000-8000 people died of this cancer every year in Taiwan. DNA microarray (DNA chip) is a very powerful tool to clarify the genetic changes in cancers. Expression profiling techniques have been used to simultaneously monitor the expression of thousands of genes from human tumor samples. It has been successfully used to predict clinical outcome and survival as well as classify different types of cancer. In this study, we will use the DNA chip to study the genetics in liver cancer patients.

DETAILED DESCRIPTION:
The clinical samples will be collected in the NTUH, while the DNA microarray works will be done in Biomedical Engineering Center (BMEC) of ITRI.

Patients A total of 40 cases of HCC patients (20 HBV-related HCC and 20 HCV-related HCC) who received surgical resection in National Taiwan University Hospital will be enrolled from our tissue banks. The diagnosis of HCC was confirmed by pathological examination. The surgical specimens were frozen immediately after surgery and stored in -140°C. The clinicopathological data will be retrospectively obtained from chart reviews.

Another total of 40 new HCC patients who receive surgical resection in National Taiwan University Hospital will be collected. The healthy subjects and patients chronically infected with HBV or HCV without HCC will be used as controls. The whole bloods will be collected before, one and six months after operation. The diagnosis of HCC will be confirmed by pathology. In addition to the whole bloods, the surgical specimens will be frozen immediately after surgery and stored in -140°C.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma

Exclusion Criteria:

* multiple cancers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan